CLINICAL TRIAL: NCT00259545
Title: Prospektive, Randomisierte Doppelblinde Studie Zur Wirksamkeit Von Intestinal Retardiert Freigesetztem Phosphatidylcholine Bei therapierefraktärer Colitis Ulcerosa Mit Chronisch Aktivem Verlauf Unter Corticosteroiden
Brief Title: Retarded Phosphatidylcholine in Steroid-Dependent Chronic Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Professor Wolfgang Stremmel (Unknown); Dietmar Hopp Stiftung (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC2; EC - L71/2003; BFARM - 402 29 17
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Ulcerative Colitis; Phosphatidylcholine
Keywords: retarded phosphatidylcholine; chronic active; steroid
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Retarded Release Phosphatidylcholine (rPC)

SUMMARY:
The purpose of this study is to evaluate if retarded release phosphatidylcholine is an effective alternative to steroid dependent or -refractory course in chronic active ulcerative colitis.

The hypothesis is, that ulcerative colitis is caused by a barrier defect of the colonic mucus layer. The background of the study is the finding, that the phosophatidylcholine content of the colonic mucus is strongly reduced in ulcerative colitis (UC) compared to healthy controls and patients with Crohn´s disease. The content was measured in non-inflamed areas of the colon in UC. Thus, we evaluate whether a substitution of colonic PC is an effective method for steroid dependent UC. See: Gut. 2005 Jul;54(7):966-71. Stremmel et al.

DETAILED DESCRIPTION:
Design: Prospective, randomized, placebo-controlled, double-blinded study.

Population: 60 patients with chronic active ulcerative colitis and steroid dependency

Inclusion: Chronic active ulcerative colitis, clinical index 5 or more, endoscopic Index 5 or more, steroid dependent course since at least 4 months.

Main criteria: complete steroid reduction

ELIGIBILITY:
Inclusion Criteria:

* Signed Letter of Content
* diagnosis of ulcerative colitis (clinical, endoscopic and histologic evidence)
* chronic active and steroid dependent course over at least 4 months (CAI > 4, EAI > 4)

Exclusion Criteria:

* infectious colitis
* toxic megacolon
* ulcerative proctitis or less than 20cm inflamed

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-02; Study Completion 2006-02

PRIMARY OUTCOMES:
complete steroid reduction

SECONDARY OUTCOMES:
remission, life quality, clinical indices, endoscopic indices, histological score, subgroup analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Stremmel, Professor, Principal Investigator — Heidelberg University
Locations (1):
- University Heidelberg - Medical Department 4 - Gastroenterology, Heidelberg, Germany

REFERENCES:
- [Background] Stremmel W, Merle U, Zahn A, Autschbach F, Hinz U, Ehehalt R. Retarded release phosphatidylcholine benefits patients with chronic active ulcerative colitis. Gut. 2005 Jul;54(7):966-71. doi: 10.1136/gut.2004.052316. PMID 15951544
- [Derived] Stremmel W, Ehehalt R, Autschbach F, Karner M. Phosphatidylcholine for steroid-refractory chronic ulcerative colitis: a randomized trial. Ann Intern Med. 2007 Nov 6;147(9):603-10. doi: 10.7326/0003-4819-147-9-200711060-00004. PMID 17975182